CLINICAL TRIAL: NCT01748019
Title: Phase I Dose Finding and Pharmacokinetic Study of the Intravenous Camptothecin ST1968 in Patients With Solid Tumors
Brief Title: ST1968 Intravenous (Weekly) in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: Southern Europe New Drug Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST1968-DM-06-001
Record Dates: First submitted 2012-06-12; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-06

CONDITIONS: Solid Tumors
Keywords: ST1968; Camptothecin; Solid tumors; Topoisomerase I
MeSH Terms: interventions — namitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ST1968 (Experimental): ST1968 once a week for 2 weeks every 3 weeks (protocol amendment: once every 3 weeks
  --------------------------------------------------------------------------------
  Interventions: Drug: ST1968

INTERVENTIONS:
Drug: ST1968 — ST1968 once a week for 2 weeks every 3 weeks (protocol amendment: once every 3 weeks
  Other Names: Namitecan

SUMMARY:
ST1968 is a novel camptothecin derivative which interacts with topoisomerase I-DNA complex, inducing S-Phase specific cytotoxicity. It is endowed with a potent antitumor activity and an increased Therapeutic Index with respect to the clinically used analogues (i.e.irinotecan and topotecan) in some xenograft models (ovary, colon, head & neck, cervix). Anti-tumor activity has been also noted in platinum resistant ovarian cell xenografts and in topoisomerase I mutant prostate cell lines. The acceptable toxicity profile in animals and the activity in camptothecin-resistant cell lines make ST1968 a good candidate for clinical trials.

DETAILED DESCRIPTION:
Multicenter, open label, uncontrolled Phase I pharmacokinetic trial to determine the Maximum Tolerated Dose (MTD) of ST1968 given intravenously (I.V.) once every week for 2 consecutive weeks every 3 weeks and the MTD of ST1968 given I.V. once every 3 weeks. A starting dose of 1.5mg/m2 given as a flat dose of 2.5mg is defined, given once on Day 1, Day 8 every 21 Days (D1, D8 Q21D schedule), over 2 h. Starting dose for the Day 1 every 21 Days (D1 Q21D schedule) has to be determined from the MTD of D1, D8 Q21D schedule.

Plasma, urine pharmacokinetics in all patients (minimum of 3 pts for each cohort) during the first cycle of treatment and in at least 6 patients at the Recommended Dose (RD).

During the study any hints of anti-tumor activity will also be evaluated by RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of solid tumors for which therapy of proven efficacy does not exist.
* Preferably measurable disease
* ECOG performance status ≤ 1.
* Age ≥ 18 years.
* Ongoing toxicity associated with prior anticancer therapy ≤ grade 1 (NCI-CTCAE V3.0).
* Maximum of 2 prior chemotherapy lines for advanced disease (not including neoadjuvant or adjuvant chemotherapy)
* Adequate hematological, liver and renal function
* Hemoglobin ≥ 9 g/dl; ANC ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L;
* Serum bilirubin ≤ upper normal limit (UNL). ALT, AST ≤ UNL but ≤ 2.5 x UNL in case of liver metastases; alkaline phosphatase (liver isoenzyme fraction) ≤ UNL or ≤ 1.5xULN in case of liver metastases; albumin within normal limits;
* Creatinine ≤1.5 mg/dl or calculated creatinine clearance ≥ 60 ml/min.
* Life expectancy of at least 3 months
* Capacity of understanding the nature of the trial and giving written informed consent.

Exclusion Criteria:

* Less than 4 weeks since last chemotherapy, radiotherapy or prior investigational therapy. Less than 2 weeks since last hormone or immunotherapy or signal transduction therapy.
* Active infection.
* Presence of cirrhosis or chronic hepatitis
* Presence of serious cardiac (congestive heart failure, angina pectoris, myocardial infarction within one year prior to study entry, uncontrolled hypertension or arrhythmia), neurological or psychiatric disorder.
* Presence of uncontrolled intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
* Symptomatic brain metastases (this does not include primary brain tumors) or leptomeningeal disease.
* Pregnancy or lactation or unwillingness to use adequate method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ST1968 given I.V. once every week for 2 consecutive weeks every 3 weeks and MTD of ST1968 given I.V. once every 3 weeks | 21 days
  2/6 patients with a Dose Limiting Toxicity (DLT) at the first cycle (21 days)

SECONDARY OUTCOMES:
Adverse events, physical examination and laboratory tests (hematology and biochemistry) as a measure of safety and tolerability | 21 days of each cycle of therapy
  safety assessments (routine physical examinations and laboratory evaluations) and severity of adverse events based on the NCI-Common Terminology Criteria for Adverse Events V. 3.0 (NCI-CTCAE)
Tumor response | 4 weeks
  objective tumor response based on RECIST criteria
Tmax, Cmax, AUC0-24, AUC-last, T1/2,CL | 21 days
  full blood and urine PK

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Hess, MD, Study Chair — Kantonsspital St. Gallen, 9700 St. Gallen - Switzerland